CLINICAL TRIAL: NCT00218504
Title: Cue Reactivity Model for Assessing Pharmacologic Intervention in Treatment of Cannabis Use Disorders (Study 2)
Brief Title: Responses to Marijuana-Related Cues Versus Neutral Cues in Adults Taking Tetrahydrocannabinol (THC) - 2
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Leslie Lundahl, Principal Investigator, Wayne State University
Other Study IDs: NIDA-19236-2; R21DA019236 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Tetrahydrocannabinol — Participants will be randomly assigned to receive an oral dose of 10 mg of THC, 20 mg of THC, or placebo.

SUMMARY:
The majority of past research on marijuana treatment has targeted the alleviation of withdrawal symptoms. Minimal focus has been placed on how altering craving effects may play a role in treating marijuana addiction. Treatment with tetrahydrocannabinol (THC), the main ingredient in marijuana responsible for its reinforcing effects, may decrease marijuana cravings. The purpose of this study is to evaluate the effect of THC pre-treatment on responses to marijuana-related cues versus non marijuana-related cues in individuals addicted to marijuana.

DETAILED DESCRIPTION:
Marijuana is the most commonly used illegal drug in the United States; more than 2 million Americans either abuse or are dependent on the drug. Therefore, there is a clear need for treatment options. Past research on marijuana treatments has focused on alleviating withdrawal symptoms. Minimal focus has been placed on how altering craving effects may play a role in treating marijuana addiction. Treatment with THC, a component of marijuana that causes the "high" sensation, may reduce marijuana cravings. This study will evaluate the subjective and physiological responses to marijuana-related cues versus non marijuana-related cues in marijuana users who have been pre-treated with THC.

Participants will attend three 6-hour sessions, each separated by at least 7 days. Prior to each testing session, participants will spend the night at the Psychiatric and Addiction Research Center at Detroit Receiving Hospital in order to ensure no alcohol or drug use during the 12 hours preceding the session. Participants will be randomly assigned to receive an oral dose of 10 mg of THC, 20 mg of THC, or placebo. They will then undergo a cue exposure test during which they will be shown a nature video and will be asked to handle and smell various items; these will act as neutral, non marijuana-related cues. Next, the participants will watch a video of individuals smoking marijuana and will be asked to handle and smell marijuana-related items; these will act as the marijuana-related cues. Heart rate and skin temperature will be monitored continuously throughout each session with the use of electrodes and a skin thermometer. Prior to and after the cue exposure sessions blood pressure will be measured and questionnaires will be administered to assess drug cravings as well as related mood states. Prior to leaving the clinical center, the participants' vital signs will be evaluated to ensure that any cue-related physiological changes have returned to normal. Following the end of the study session, participants will have the option of talking to a clinician experienced in dealing with drug cravings.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnosis criteria for marijuana dependence
* Able to read and write in English
* Positive urine test for marijuana
* If female, must be willing to use contraception throughout the study

Exclusion Criteria:

* Meets DSM-IV diagnosis criteria for a psychiatric illness
* History of a psychotic disorder
* Seeking treatment for marijuana dependence
* Neurologic disease, including structural brain abnormalities (e.g., neoplasms), stroke, seizures, infectious disease, head trauma resulting in unconsciousness, or evidence of neurologic illness resulting from HIV/AIDS
* Cardiovascular disease, including edema, chest pain or palpitations after exertion or drug use, myocardial infarction (heart attack), systolic blood pressure greater than 160 mm Hg or less than 95 mm Hg, or diastolic blood pressure greater than 95 mm Hg
* Pulmonary disease, including apnea, cor pulmonale, tuberculosis, dyspnea, orthopnea, or tachypnea
* Systemic disease, including endocrinopathies, kidney or liver failure, hypothyroidism, adrenocortical insufficiency, or autoimmune disease involving the central nervous system
* Currently dependent on any drug other than marijuana or nicotine
* Cognitively impaired
* Pregnant or breastfeeding

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Marijuana dependent volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2005-12; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Marijuana craving | Measured throughout the cue exposure session

CONTACTS AND LOCATIONS:
Overall Officials: Leslie H. Lundahl, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Lundahl LH, Greenwald MK. Magnitude and duration of cue-induced craving for marijuana in volunteers with cannabis use disorder. Drug Alcohol Depend. 2016 Sep 1;166:143-9. doi: 10.1016/j.drugalcdep.2016.07.004. Epub 2016 Jul 18. PMID 27436749
- [Derived] Lundahl LH, Greenwald MK. Effect of oral THC pretreatment on marijuana cue-induced responses in cannabis dependent volunteers. Drug Alcohol Depend. 2015 Apr 1;149:187-93. doi: 10.1016/j.drugalcdep.2015.01.046. Epub 2015 Feb 11. PMID 25725933